CLINICAL TRIAL: NCT00885209
Title: Evaluation of the PillCam Colon Capsule Endoscopy Preparation and Procedure
Brief Title: Evaluation of the PillCam™ Colon Capsule Endoscopy (PCCE) Preparation and Procedure
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-108
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2010-03

CONDITIONS: Colonic Diseases
Keywords: Colonic Diseases
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients that are indicated for colonoscopy, who are suspected or known to suffer from colonic diseases.

SUMMARY:
The purpose of this study is to evaluate the effect of a modified Prep and procedure on colon cleansing level and capsule excretion rate.

DETAILED DESCRIPTION:
The evaluation of subjects with suspected colonic disease includes endoscopic imaging by colonoscopy and radiologic imaging such as air-contrast barium enema, or CT colonography . The Given® Diagnostic System offers an alternative approach for endoscopic visualization of the colon using capsule endoscopy, an ingestible device which contains imagers, light sources, a power source and a RF transmitter. Advantages of the Given® Diagnostic System include the elimination of the need for sedation, the minimally invasive, painless nature of the exam, and the ability to pursue normal daily activities immediately following the procedure . Furthermore, compared to standard colonoscopy, the Given® Diagnostic System may be more readily accepted by the subjects, thereby improving subjects' willingness to undergo a diagnostic evaluation of the colon and comply with colorectal cancer screening recommendations. The PillCam™ SB capsule (formerly M2A® Capsule) that was FDA-approved in August 2001 for small bowel evaluation has been ingested to date by more than 500,000 people worldwide and is well accepted by patients and physicians as well as the processional societies. However, adequate visualization of the colon cannot be achieved with the standard PillCam™ SB capsule because of the anatomical and physiological properties of the colon which are significantly different than the small bowel. Moreover, other issues that limit the evaluation of the colonic mucosa by the standard PillCam™ SB procedure include an unsatisfactory level of colon cleanliness and slow progression of the PillCam™ SB capsule through the colon during the desired examination time. Therefore, the development and introduction of a specially designed, customized colon capsule combined with a dedicated capsule colonoscopy procedure protocol will allow for more efficient evaluation of the colonic mucosa. This is expected to improve the capability of the Given® Diagnostic System to detect colonic pathologies and to serve as a diagnostic and screening tool for colonic disease. Further details of the PillCam™ Colon Capsule Endoscope (PCCE) can be found in the device description section.

This is a pilot study that is designed to compare the levels of cleanliness and visualization of colon achieved by colon capsule endoscopy when using different regimens for preparation of the colon. Furthermore, capsule colonoscopy and colonoscopy procedures will be compared in regards to the level of colon cleanliness and detection of lesions in the colon.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:
* Subject is between the ages of 50-75 years and clinically indicated for conventional colonoscopy-
* Subject is 18-50 years of age suspected /known to suffer from colonic disease and was referred for colonoscopy for any standard indication including, but not limited to: rectal bleeding, melena, positive stool testing for occult blood, recent change of bowel habits, screening for colorectal cancer, ulcerative colitis, signs of colonic lesions on an imaging study)-
* No more than 25% of subjects (for each site) will be recruited from group B with a minimum of 20%

Exclusion Criteria:

* The presence of any of the following will exclude a subject from study enrollment:
* Subject has dysphagia or any swallowing disorder
* Subject has congestive heart failure
* Subject has high degree of renal insufficiency
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator
* Subject has a cardiac pacemaker or other implanted electromedical device.
* Subject has any allergy or other known contraindication to the medications used in the study
* Subject is not eligible for colon preparation with sodium phosphate solution due to the presence of underlying conditions according to the clinical judgment of the investigator.
* Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Subject with any condition believed to have an increased risk for capsule retention such as Crohn's disease, intestinal tumors, radiation enteritis, or NSAID enteropathy,
* Subject has any condition, which precludes compliance with study and/or device instructions.
* Women who are either pregnant or nursing at the time of screening, who intend to be during the study period, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
* Subject suffers from life threatening conditions
* Subject currently participating in another clinical study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients that are indicated for colonoscopy, who are suspected or known to suffer from colonic diseases
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Colon cleansing level score | within 7 days
Number of colon capsules excreted over time | within 7 days

SECONDARY OUTCOMES:
Accuracy parameters of PCCE, compared to colonoscopy. | within 7 days
Diagnostic yield of PCCE compared to standard colonoscopy | within 7 days
Number of complete capsule procedure | within 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Munoz, Prof. Dr., Principal Investigator — Clinica Universitaria de Navarra
Locations (5):
- Spain (5):
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Georio Maranon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital virgen Macarena, Seville